CLINICAL TRIAL: NCT03237689
Title: Effects of Glucocorticoids on Cognition in HIV-infected Women
Acronym: MsSCORE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00145327; R01MH113512 (NIH)
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: The design is a two-phase study of HIV+ women who: 1) first participate in a double-blind, placebo-controlled cross-over study of a single, low dose (10 mg) of hydrocortisone versus placebo on cognition; and 2) then participate in a mechanistic, randomized, double-blind, placebo controlled trial of daily LDH for 4 weeks on cognition and side effects.
  Below includes the number of arms for the second study phase and is the phase of the study being considered a Phase 0 clinical trial. All information to follow will pertain to this phase of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only entity knowledgeable of randomization is the Johns Hopkins University Investigational Drug Service Pharmacy. They are responsible for randomizing and encapsulating the drug and placebo tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone (Experimental): Low dose hydrocortisone (10mg orally)
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Placebo tablets, made of starch 1500 powder
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Hydrocortisone — Low dose hydrocortisone (10mg)
  Arms: Hydrocortisone
Drug: Placebo Oral Tablet — capsules of starch 1500 powder
  Arms: Placebo

SUMMARY:
Despite treatment with antiretroviral therapy, women living with HIV continue to experience cognitive impairment. Psychological risk factors, including stress, impair cognition more in HIV-infected women than HIV-uninfected women. This study plans to examine a novel intervention for cognitive dysfunction that targets the mechanisms by which stress negatively affects cognitive functioning.

DETAILED DESCRIPTION:
The overall aim of this study is to contribute important foundational knowledge of the utility of targeting neuroinflammation and the hypothalamic-pituitary-adrenal (HPA) axis to improve cognition in HIV and will provide key clinical insights into the mechanisms underlying any cognitive benefit. The investigators are conducting a single-dose study of low dose hydrocortisone (LDH) followed by a 4-week study of daily LDH as a probe of the mechanisms of neuroinflammation including myeloid-lineage cells and the HPA axis in HIV-infected (HIV+) women demonstrating cognitive dysfunction and reporting high levels of stress, trauma history, and mental health risk factors which commonly occur in this population. The use of a pharmacological challenge may aid in the identification of: 1) a putative biomarker of stress- and psychiatric disorder-related neurocognitive complications in HIV-infected women and/or 2) an adjunctive, cost-effective therapy for the treatment of cognitive deficits in HIV

The design is a two-phase study of HIV+ women who: 1) first participate in a double-blind, placebo-controlled cross-over study of a single, low dose (10 mg) of hydrocortisone versus placebo on cognition; and 2) then participate in a mechanistic, randomized, double-blind, placebo controlled trial of daily LDH for 4 weeks on cognition and side effects. The clinical trial will include 100 virally suppressed HIV+ women who show elevated stress and cognitive impairment and who represent the range of psychological risk factors characteristic of this population. Next, to understand the mechanism and broader clinical significance of LDH on cognition, investigators will conduct a 4-week randomized study of the effects of daily treatment with LDH versus placebo on cognition in HIV+ women (targeted n=80).

Women meeting enrollment criteria will complete three cognitive assessments. The first and second assessments will be embedded in the double-blind, placebo-controlled, cross-over study of a single administration of LDH versus placebo (targeted n=100). Investigators will measure cognitive performance 30 minutes and 4 hours post-dosing, because an emerging literature shows that the cognitive effects of LDH depends on timing of the assessment post-dosing. The 30-minute assessment addresses how the maximal cortisol levels following LDH affect cognition. This immediate assessment is standard in studies of stress and cognition and allows for comparisons with the broader literature. More novel and clinically important is the 4-hour assessment which occurs post-peak, when cortisol levels are more steady state and typical of the broader daily cortisol profile following LDH. The third assessment will take place after 4 weeks of treatment with LDH or placebo. That assessment addresses the clinical significance and safety of longer-term LDH treatment. Lastly, the investigators will explore glucocorticoids and inflammation and immune activation as mechanisms by which LDH might affect cognition.

Objective 1 To examine immediate and delayed effects of a single administration of LDH on cognition in HIV+ women.

Objective 2 To examine the effects of a 4-week course of daily LDH on cognition in HIV+ women.

Objective 3 To investigate potential mechanisms of LDH effects on cognition in HIV+ women.

ELIGIBILITY:
Inclusion Criteria:

* Females only;
* HIV-infected;
* Able to give informed consent;
* Able to travel to study site for study participation;
* Age between 18 and 65;
* English as a first language;
* Above-average self-reported levels of perceived stress (>14 on the perceived stress scale (PSS-10)) and/or current SCID-V diagnosis of mood and/or anxiety disorder;
* Meet criteria for HIV-associated cognitive dysfunction (based on Neurocognitive test battery and instrumental activities of daily living assessment-impairment on only 1 cognitive domain is required)
* Virally suppressed and on combination antiretroviral therapy (Plasma HIV RNA<1000cp/ml and bring in medications)

Exclusion Criteria:

* Current use of hormone-based contraceptives (birth control pills or patch);
* Currently pregnant, post-partum or lactating;
* Currently regular use of steroids;
* History of closed head injury resulting in loss of consciousness greater than 1 hour;
* History of schizophrenia or schizoaffective disorder;
* Current untreated hypertension or diabetes*;
* History of dementia or any other neurologic central nervous system (CNS) or AIDS-defining disorder;
* Positive urine toxicology screen (except marijuana) or breathalyzer and/or any evidence of acute intoxication or withdrawal.
* History of substance abuse/dependence in the past six months.

Participants who present with a heretofore untreated condition (e.g., hypertension) will be excluded; however, they may be rescreened for eligibility after receiving appropriate treatment for the condition in the course of their standard medical care (at least 6 months).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test-Revised assesses total learning | change between baseline and 28 days
  a 12-item list-learning task across 3 trials used to measure total learning. Outcome=total learning across trials (range 0-36). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Hopkins Verbal Learning Test-Revised assesses verbal memory | change between baseline and 28 days
  following the 3 learning trials there is a 20-25 minute delay. After the delay, participants are asked to recall as many words as they can from the initial learning list. Outcome=delayed free recall (range 0-12).Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Wechsler Adult Intelligence Scale IV Letter-Number Sequencing assesses working memory condition | change between baseline and 28 days
  participants hear a series of letters and numbers, and then recite them back in ascending order, with the numbers first and then the letters. Outcome=total correct (range 0-24). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Line Orientation Task assesses visuospatial abilities | change between baseline and 28 days
  In each of 10 trials, a visual array of 13 lines fans out from a common point of origin. Two target lines are shown beneath each array, and participants must identify the lines within the array that match each of the two target lines. Outcome=Total correct (range=0-20).

SECONDARY OUTCOMES:
Trail Making Test Part A assesses processing speed/attention | change between baseline and 28 days
  25 circles distributed over a sheet of paper. The circles are numbered 1 - 25 and the participant should draw lines to connect the numbers in ascending order. Outcome=Time to completion (range: 10 to 300 seconds). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Trail Making Test Part B assesses mental flexibility | change between baseline and 28 days
  25 circles are distributed over a sheet of paper. Circles include both numbers (1 - 13) and letters (A - L). The participant draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). Outcome=time to completion (range: 18-300). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Comalli Stroop Test, Trial 1 assesses processing speed/attention | change between baseline and 28 days
  Participants identify aloud the colors of a series of squares. Outcome=time to completion (range: 30 to 240). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Comalli Stroop Test, Trial 2 assesses processing speed/attention | change between baseline and 28 days
  Participants read a series of color names printed in black ink. Outcome=time to completion (range: 30 to 240). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Comalli Stroop Test, Trial 3 assesses behavioral inhibition | change between baseline and 28 days
  Participants name the color of the ink but ignore the word. Outcome=time to completion (range: 50 to 240). Neuropsychological measures are normed on populations and therefore the clinical significance of a score can be assessed in relation to expected levels of performance.
Liver function as assessed by aspartate aminotransferase (AST) levels | change between baseline and 28 days
  levels from blood. Clinical significance will be determined using the Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events.
Liver function as assessed by alanine transaminase (ALT) levels | change between baseline and 28 days
  levels from blood. Clinical significance will be determined using the Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events.
Liver function as assessed by alkaline phosphatase levels | change between baseline and 28 days
  levels from blood. Clinical significance will be determined using the Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events.
renal function assessed by creatinine levels | change between baseline and 28 days
  levels from blood. Clinical significance will be determined using the Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events.
metabolic function assessed by glucose levels | change between baseline and 28 days
  levels from blood. Clinical significance will be determined using the Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events.
metabolic function assessed by hemoglobin A1c (HbA1c) | change between baseline and 28 days
  levels from blood. Clinical significance will be determined using the Division of AIDS (DAIDS) Table for grading the severity of adult and pediatric adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Leah Rubin, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Brief Report: Low-Dose Hydrocortisone Has Acute Enhancing Effects on Verbal Learning in HIV-Infected Men — https://www.ncbi.nlm.nih.gov/pubmed/28141781
- See also: Elevated stress is associated with prefrontal cortex dysfunction during a verbal memory task in women with HIV — https://www.ncbi.nlm.nih.gov/pubmed/27094924
- See also: Prefrontal cortical volume loss is associated with stress-related deficits in verbal learning and memory in HIV-infected women — https://www.ncbi.nlm.nih.gov/pubmed/26408051
- See also: Post-traumatic stress is associated with verbal learning, memory, and psychomotor speed in HIV-infected and HIV-uninfected women — https://www.ncbi.nlm.nih.gov/pubmed/26404435
- See also: The association of perceived stress and verbal memory is greater in HIV-infected versus HIV-uninfected women — https://www.ncbi.nlm.nih.gov/pubmed/25791344